CLINICAL TRIAL: NCT01283243
Title: Prospective Study for Assessment of Normal Value of Acoustic Radiation Force Impulse (ARFI) Elastography in HIV Patients Without Abnormal Liver Function and Chronic Liver Disease
Brief Title: Assessment of Normal Value of Acoustic Radiation Force Impulse (ARFI) Elastography in HIV Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Collaborators: Severance Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2010-0027
Record Dates: First submitted 2011-01-21; First posted 2011-01-25 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: HIV Infection
Keywords: ARFI Imaging; Normal values; HIV infection
MeSH Terms: conditions — HIV Infections | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HIV patients with normal liver status: HIV patients without abnormal liver function and chronic liver disease
  Interventions: Device: Acoustic radiation force impulse imaging

INTERVENTIONS:
Device: Acoustic radiation force impulse imaging — Acoustic radiation force impulse (ARFI) imaging were measured 10 times in each patient.The region of interest was chosen in an area where the normal liver parenchyma was at least 6 cm thick and free of large blood vessels was chosen. A measurement depth of 2 cm below the liver capsule was chosen to standardize the examination.
  Other Names: ARFI imaging

SUMMARY:
This is a prospective cohort single center study for assessment of normal value of acoustic radiation force impulse elastography and fibroscan in HIV patients without abnormal liver function and chronic liver disease.

DETAILED DESCRIPTION:
HIV positive patients who have liver dysfunction have shown to be correlated with high mortality and morbidity. To date, ARFI elastography has been known to correlate with the degree of liver fibrosis in chronic liver disease. However, ARFI velocity has not yet been reported in HIV patients. The aim of this study was to identify the normal range of ARFI velocity and liver stiffness value by recruiting HIV patients without abnormal liver function and chronic liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Age > 20 years
* HIV positive patients
* The patients who is willing and able to provide written informed consent to participate in this study

Exclusion Criteria:

* Co-infected with HIV and HBV or HCV
* History of any other forms of liver disease
* Any gross abnormality on the imaging finding including MRI and CT
* Any laboratory abnormalities regarding liver condition (Platelet count < 150 x 103/ul, Fasting glucose > 110 mg/dl, AST > 40 IU/L, ALT> 40 IU/L, Albumin < 3.3 g/dl, Total bilirubin > 1.2 mg/dl, GGT> 54 IU/L, ALP > 115 IU/L , Ferritin > 322 ng/ml)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV patients without abnormal liver function and chronic liver disease
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of ARFI velocity in HIV patients | 2 years
  Measurement of ARFI velocity is non-invsive ultrasonographic technique. It is performed with a abdominal convex probe which is same probe as conventional ultrasonography. Short-duration acoustic radiation forces result in shear-wave propagation away from the region of excitation and are tracked using ultrasonic correlation-based methods. This results are called ARFI velocity which is expressed as meters per second

CONTACTS AND LOCATIONS:
Overall Officials: Kwang-Hyub Han, MD, Study Chair — Yonsei University Colleage of Medicine; Seung Up Kim, MD, Principal Investigator — Yonsei University Colleage of Medicine
Locations (1):
- Severance Hospital, Seoul, South Korea